CLINICAL TRIAL: NCT00878605
Title: Development of A Novel Anti-Hyperglycemic Agent
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to reach accrual target.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-010-08F
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Diabetes
Keywords: Diabetes; Cyclo-Z
MeSH Terms: conditions — Diabetes Mellitus | interventions — Z 008; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cyclo-Z (minimally effective) (Experimental): 3mg CHP plus 20mg zinc containing gel capsule;
  Interventions: Drug: Cyclo-Z
- Cyclo-Z (maximally effective) (Experimental): 9mg CHP plus 20mg zinc containing gel capsule;
  Interventions: Drug: Cyclo-Z
- Cyclo-Z (not additionally effective) (Experimental): 15mg CHP plus 20mg zinc containing gel capsule
  Interventions: Drug: Cyclo-Z
- Placebo (for CHP) (Placebo Comparator): Placebo capsules containing no zinc or CHP
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclo-Z — Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
  Other Names: CHP
  Arms: Cyclo-Z (maximally effective); Cyclo-Z (minimally effective); Cyclo-Z (not additionally effective)
Drug: Placebo — Placebo control
  Other Names: Sugar pill manufactured to mimic Cyclo-Z
  Arms: Placebo (for CHP)

SUMMARY:
The purpose of this clinical trial is to test the effectiveness and safety of a new anti-diabetes drug (Cyclo-Z) for the prevention and treatment of Type 2 diabetes. This study will determine dose-dependent efficacy and safety of this new drug for the treatment of human diabetes. The Food and Drug Administration has granted approval for the use of this investigational product to be used in a study [FDA approval (Investigational New Drug) IND #: 61,897]. This new drug is thought to work by increasing the amount of zinc in your body, which in turn should improve your sugar metabolism. If this study successfully proves that Cyclo-Z is effective for the treatment of diabetes and is without significant side effects, a large, multi-center study of diabetic patients will then be performed.

DETAILED DESCRIPTION:
We have demonstrated that a cyclic dipeptide Cyclo (his-pro) plus zinc (Cyclo-Z) treatment improved clinical conditions of diabetes in various animal models and a phase 1 clinical trial. The main objective of this study is to demonstrate that this product is safe and effective for the treatment of human diabetes.

Research Plan This is a randomized, double blinded, placebo-controlled, and parallel study. In this study, we will recruit 120 hypoglycemic drug na ve type 2 diabetic patients and randomize them into 4 groups of 30 subjects each to compare the effects of a Cyclo-Z capsule containing Cyclo-His Pro (CHP) 0 (placebo), 3 mg (minimally effective), 9 mg (optimally effective), or 15 mg (no-additional effect) plus 20 mg zinc on diabetic symptoms in a 12-week trial period. The primary outcome of this study is improvement of hemoglobin A1c; secondary outcomes are fasting blood glucose, 2 hours postprandial glucose and glucose tolerance test. Safety will be assessed by the presence of severe adverse events (SAEs), adverse events (AEs), any changes of vital signs, physical exams, blood hematology, chemistry, liver, renal, thyroid function tests, urine analysis and zinc, copper levels.

Clinical Significance The proposed study has a direct impact on veteran's healthcare service. The applicant has obtained two types of US and international patent approvals for preventing and treating human diabetes and obesity with Cyclo-Z. One patent application for Alzheimer's disease treatment has just been approved. These patent rights are now assigned to the DVA. Based on our background studies and observation we anticipate the proposed Phase 2a clinical trials will prove that Cyclo-Z treatment is safe and effective for the treatment of human diabetes and we will be able to present a new class of anti-diabetes drug to improve healthcare of both the VA diabetic patients and the general public.

ELIGIBILITY:
Inclusion Criteria:

1. History of type 2 diabetes mellitus who are na ve to hypoglycemic treatment, inadequately controlled by diet and exercise alone or oral medications.
2. Hemoglobin A1c level of 6.5 % to 8.0 % inclusive. Subjects not taking hypoglycemic drugs with HgbA1c of 6.0% to 6.5% must have a diagnosis of Diabetes Mellitus (DM).
3. Fasting blood glucose levels reasonably stable for at least 2 months or during the two-week lead-in-period.
4. Ethnicity: All ethnic groups.
5. Gender: Both men and women.
6. Female with reproductive potential must not be pregnant or lactating, and using reliable contraception methods.
7. Age >18 years old.

Exclusion Criteria:

1. Taking insulin.
2. History of diabetic ketoacidosis or hyper osmolar non-ketotic coma.
3. Diabetes Mellitus related end-organ damage:

   * Evidence of diabetic autonomic and peripheral neuropathy
   * Diabetic proliferative retinopathy, based on eye exam by ophthalmologist
   * Diabetes nephropathy defined by > 500 mg/24 hour urinary albumin excretion
4. Any disease likely to limit life span and/or increase risks of interventions:

   * Screening carotid B-mode ultrasound indicating clinically significant stenos in the common carotid arteries requiring intervention by angioplasty or resection.
   * Cancer treatment in the past 5 years, with the exception of cancers that have been cured, and carry a good prognosis.
   * Infectious disease: HIV positivity, active tuberculosis, or pneumonia.
5. Cardiovascular disease:

   * Hospitalization for treatment of heart disease in the past 12 months.
   * New York Heart Association Functional Class > 2.
   * Left Bundle branch block on EKG.
   * Third degree atrioventricular block on EKG.
   * Uncontrolled hypertension with average systolic blood pressure of > 160 mmHg on two screening visits and diastolic blood pressure > 95 mmHg on two screening visit.
   * Pulse rate > 95 beats per minute on both screening visits.
   * Stroke or transient ischemic attack in the past 12 months.
6. Gastrointestinal disease:

   * Chronic hepatitis or cirrhosis.
   * Episode of alcoholic hepatitis or alcoholic pancreatitis.
   * Inflammatory bowel disease requiring treatment in the past 12 months.
   * Recent or significant abdominal surgery (e.g. gastrectomy, gastric bypass).
7. Renal disease: Serum creatinine > 1.5 mg/dL for men, and > 1.4 mg/dL for women.
8. Lung disease:

   * Chronic obstructive airway disease or asthma requiring daily therapy.
   * Use of home oxygen.
9. Anemia: Hematocrit of < 36.0% in men or < 33% in women.
10. Conditions or behaviors likely to affect the conduct of the study

    * Unable or unwilling to give informed consent.
    * Unable to communicate with the clinic staff.
    * Unwilling to accept treatment assignment by randomization.
    * Weight loss of > 10% in the past 6 months.
    * Unable to walk without any assisted device.
    * Major psychiatric disorder which would impede conduct of the research.
    * Excessive alcohol intake (more than 2 drinks/day)
11. Medications

    * Psychoactive agents such as Monoamine oxidase inhibitors and Antidepressive agents (lithium, prozac, zoloft, serzone, paxil, effexor)
    * Systemic use of glucocorticoids steroids within previous 6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment commenced on June 1, 2009 under version 1.0 of the protocol, upon approval of the study by the IRB. The first participant was enrolled April 2010, and the last January 2013. Participants received either Cyclo-Z gel 3mg + 20mg zinc; Cyclo-Z gel 9 mg + 20mg zinc; Cyclo-Z gel 15mg + 20mg zinc or Placebo once daily for 12 weeks.
Groups:
- Arm 1: Placebo control
  Placebo: Placebo control
  Participants received placebo tablet orally daily for 12 weeks.
- Arm 2: Active medication
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
  Participants received Cyclo-Z gel 3mg + 20 mg zinc orally per day for 12 weeks.
- Arm 3: Active medication efficacy dose
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
  Participants received Cyclo-Z gel 9mg + 20 mg zinc orally per day for 12 weeks.
- Arm 4: Active medication high dose
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
  Participants received Cyclo-Z gel 15mg + 20 mg zinc orally per day for 12 weeks.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 10 | 10 | 9 | 9
Completed | 7 | 7 | 8 | 6
Not Completed | 3 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cyclo-Z Gel 3mg + 20 mg Zinc: Active medication
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
- Cyclo-Z Gel 9mg + 20 mg Zinc: Active medication efficacy dose
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
- Cyclo-Z Gel 15mg + 20 mg Zinc: Active medication high dose
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
- Total: Total of all reporting groups
Arm/Group | Placebo | Cyclo-Z Gel 3mg + 20 mg Zinc | Cyclo-Z Gel 9mg + 20 mg Zinc | Cyclo-Z Gel 15mg + 20 mg Zinc | Total
Number analyzed (Participants) | 10 | 10 | 9 | 9 | 38
Age, Continuous [Mean (Full Range); unit: years] | 58.7 [18 to 80] | 61.9 [18 to 80] | 63.4 [18 to 80] | 59.5 [18 to 80] | 60.8 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 3 | 5
  Male | 9 | 9 | 9 | 6 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 9 | 9 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 8 | 8 | 29
  White | 2 | 4 | 1 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Demographics [Number; unit: participants] | 10 | 10 | 9 | 9 | 38

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C
Description: % change HgbA1c from baseline to 12 weeks.
Time Frame: Baseline and Week 12
Arm/Group | Placebo | Cyclo-Z Gel 3mg + 20 mg Zinc | Cyclo-Z Gel 9mg + 20 mg Zinc | Cyclo-Z Gel 15mg + 20 mg Zinc
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Arm 1: Placebo control
  Placebo: Placebo control
- Arm 2: Active medication
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
- Arm 3: Active medication efficacy dose
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
- Arm 4: Active medication high dose
  Cyclo-Z: Cyclo-Z is a cyclic dipeptide Cyclo (his-pro) plus zinc that may lower blood glucose
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/9 | 1/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=10) | Arm 2 (N=10) | Arm 3 (N=9) | Arm 4 (N=9)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=10) | Arm 2 (N=10) | Arm 3 (N=9) | Arm 4 (N=9)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic Reaction to Shellfish (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This subject was terminated early and data was not analyzed due to inability to recruit and therefore small numbers of subjects to analyze leading to uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes